# **Informed Consent**

"Empowerment Self-Defense Training for the Prevention of Victimization of Transgender Women" ID: R21MD014807 NCT04934189 3/30/2021



## **Participant ID**



## **Study Consent:**

## **Participant ID**

Please enter the last 4 digits of your phone number, followed by the first initial of your first name.

For example, if my name was Jane and my phone number was (000) 123-4567, I would enter

This will be your participant ID. You will be asked to provide this ID throughout your participation in the study.

#### Consent

THE CITY UNIVERSITY OF NEW YORK **Hunter College Department of Psychology** 

INTERNET BASED INFORMED CONSENT

Title of Research Study: Empowerment Self-Defense Training for the Prevention of Violence among Transgender Women (Phase 2)



Principal Investigator: Dr. Danielle Berke, PhD

**Assistant Professor of Psychology** 

You are being invited to participate in this research study because you are an English-speaking trans woman or trans femme, are over the age of 18, and have expressed interest in participating in an empowerment self-defense program. The purpose of this research study is to tailor an empowerment self-defense program for the prevention of violence among trans women and trans femmes.

Participation in this research is voluntary. If you agree to participate, we will ask you to participate in an in-person Empowerment Self-Defense course. The course will involve five four-hour sessions occurring each Sunday for five consecutive weeks. You will be asked to complete a brief online survey before the first day of the course, after the last day, and 6 months after completing the course. Additionally, after each of the five course sessions you will be asked to complete a very brief evaluation of the session. We will also have an exit interview completed remotely over Zoom once you have completed the course. During each course session, you will learn physical and verbal skills tailored for the prevention of violence faced by trans women and trans femmes. You will also complete a series of online questionnaires about your behaviors, experiences, thoughts and emotions.

It is important for you to know that while your consent is for the full study, including the Empowerment Self-Defense course and the study questionnaires, if you later decide to withdraw from the study questionnaires you will still be able to participate in the Empowerment Self-Defense course. Similarly, if you consent to participate in this research study but later decide to drop out of the Empowerment Self-Defense course, you will still be able to participate in the questionnaires. Compensation, however, will only be distributed after the completion of each questionnaire.

#### **Study Payment:**

- You can earn up to \$180 in Amazon gift cards for survey completion, and up to \$50 in cash for self-defense session evaluations.
- After each online questionnaire (approximately 30 minutes each), we will send a gift card to your email, and after the third and fifth self-defense session, we will compensate you in cash in-person, \$10 for each class evaluation form completed (approximately 2 minutes each) (one per class) for a total of \$50.
- Payment for the study surveys increases over time: You will receive \$40 for the baseline survey, \$30 for the follow-up survey after the course and \$30 for the exit interview after the course (approximately 30 minutes), and \$80 for the 6-month follow-up survey.

This study does not pose any significant risk for participating beyond minimal discomfort or anxiety from the discussion of personal or emotional topics. You may be uncomfortable answering some of the questions. If you are bothered by any of the questions, you may skip any question you do not wish to answer or withdraw from the study without penalty. If you choose to withdraw after study procedures, if it is within 14 days of the interview session all study data (including the audio recording) will be permanently deleted. Beyond 14 days from the interview session, if you choose to withdraw consent, your data cannot be erased.

If you feel that you no longer want to complete the empowerment self-defense course, surveys, or the exit interview, you may take a break or completely stop at any time. You will not benefit directly from participation in this research, but your participation may help inform the development of interventions to prevent violent victimization and will potentially benefit the health and safety of the greater trans femme community.

To ensure the accuracy of our findings, audio recording files will be stored for later transcription and review by the research team. Thus, we are requesting your permission to video-record the interview session. If you would like a personal copy of the interview recording, you can request one before or after your interview and we will provide you with a secure link that will take you to a downloadable copy. You will have one week to use the link to download the recording. If you do not

#### **Qualtrics Survey Software**



wish to have a personal copy of the recording or the seven day window for downloading has passed, the digital video recording file will be deleted immediately and will not be saved or stored. The audio-only file will be saved for transcription. You have the right to delete the audiorecording after the interview. If you would like to erase the audio-recording, you will be asked to contact the lab within 14 days of the completion of your interview session in order to do so.

### **Confidentiality:**

We will make our best efforts to maintain confidentiality of any information that is collected during this research study, and that can identify you. We will disclose this information only with your permission or as required by law.

We will protect your confidentiality by the use of the following methods:

- Your responses will remain confidential. All identifiable information will be removed from the questionnaire data collected. Participant consent forms will be stored separately from the study data, so that the study data will be collected using only a unique participant ID number, and are not identifiable by participant name. The assigned participant ID number will be used to link study responses and audio recordings to one another.
- Hard copies of interview answer sheets, questionnaires, and any other files containing participant ID numbers will be stored in a locked file cabinet in the Pl's locked laboratory. Electronic copies of study data will be stored on an online password-protected, backed up lab server that is accessible only by lab personnel.
- The labels on these files will constitute a link between identifiable information (i.e., audio recording) and your participant ID number, which will be used to link other study data together.
- The video recordings will be recorded using the secure Zoom online video conferencing platform. Following the interview, if requested, you will be given a secure link to access and download a personnal copy of the recording. If you do not wish to obtain a copy or the seven day window for download has passed, the video recording file will be immediately deleted and will not be saved or stored. The audio-only file will be downloaded from Zoom onto the local desktop and re-uploaded to a secure password protected lab drive. The local desktop copy will be immediately deleted following upload to the secure lab drive.
- · You have the right to erase the audio recording after the interview. If you would like to delete the audio recording, you will be asked to contact the lab within 14 days of the completion of your session in order to do so. The audio-only file labeled with your participant ID number will be saved for transcription, and will contain your voice but will not contain your name.
- The audio recordings will be transcribed verbatim to facilitate qualitative analysis of core themes. These themes, in turn, will be used to inform the development of a culturally tailored violence prevention intervention for transwomen. Any identifying information will be omitted during the transcription process. Only members of the study team will be able to access the audio recordings taken during the lab session. Your responses will remain confidential.
- · Study data include some demographic information, so identification at the level of race/ethnicity or age is possible.
- We will securely retain data (including original audio recordings) for three years, then destroy
- Study data will not be stored or distributed for future research studies.

The research team, authorized CUNY staff, and government agencies that oversee this type of research may have access to research data and records in order to monitor the research. Publications and/or presentations that result from this study will not identify you by name.

Your participation in this research is voluntary. If you have any questions, you can contact Dr. Danielle Berke, Principal Investigator, by phone at 201-844-8068 or by email at BerkeLab@hunter.cuny.edu. If you have any questions about your rights as a research participant or if you would like to talk to someone other than the researchers, you can contact CUNY Research Compliance Administrator at 646-664-8918 or HRPP@cuny.edu.



| If you agree to be video-recorded during the interview as part of this research study, please select "Yes, I consent to being video-recorded as part of this research study" below. |
|---|
| I agree to be video-recorded during the interview, with the understanding that I can request a personal copy of the recording, which I will have one week following the interview to download. If I do not request a copy, or do not download it within 7 days I understand that this video recording will be deleted immediately. I understand that I have the right to erase the audio recording taken as part of this research. If I would like to delete the audio recording, I will contact the lab within 14 days of the completion of my interview session in order to do so. |
| Please indicate below whether you would permit the researchers to contact you in the future for participation in other research studies. |
| I agree to be contacted in the future for further participation in this and other research studies. I do not agree to be contacted in the future for further participation in this and other research studies. studies. |
| If you agree to participate in this research study, please select "Yes, I have read and understood the procedures and risks involved in the research study. I consent to participate in the research study" below. |
| Yes, I have read and understood the procedures and risks involved in the research study. I consent to participate in the research study. |
| Powered by Qualtrics |